CLINICAL TRIAL: NCT04235543
Title: Occurrence of Traumatic Dental Injury in a Group of Egyptian Autistic Children Compared to Normal Children: (A Cohort Study)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, marwa mousa mohamed borham, principle investigator, Cairo University
Other Study IDs: Cairo University Egypt
Record Dates: First submitted 2020-01-16; First posted 2020-01-22 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Traumatic Dental Injury; Autism Spectrum Disorder; Dental Trauma
Keywords: Autism; traumatized teeth in autistic children; occurrence of dental trauma
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- autistic children aged 6:12 years: show the occurrance of traumatic dental injury compared to normal children
- normal children aged 6:12 years: show the occurrance of traumatic dental injury

SUMMARY:
The aim of the study is to assess the occurrence of traumatic dental Injury in a group of Egyptian Autistic Children compared to normal children.

Population: Egyptian children Exposure: Autistic children. Control: Normal children. Outcome: Primary Outcome: occurence of Traumatic injury. Secondary Outcome: Risk factor, Oral habits.

DETAILED DESCRIPTION:
This study is a cohort study, the study group compromise a group of children with ASD, the control group compromise a group of normal children.

Study group will be recruited from Abbaseya Mental Health Hospital and Advance Center For Handicapped and Autistic Children.

Control group will be recruited from Diagnosis Clinic of Pediatric Dentistry and Dental Public Health Department at Faculty of Dentistry Cairo University.

The investigator will make an interview with the Parents of both groups to fill the A questionnaire (taken from different articles, modified by the investigator to accommodate the aims of the study.) then they will be assigned Informed consent, children whose parents agreed to participate in the study were recruited.

Inclusion criteria:

* Autistic and normal children.
* children aged from 6 to 12 years old irrespective of sex.

Exclusion criteria:

* Behavior of the child is inadequate.
* Children with dental structural defect.
* parents that refused to give informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Autistic and normal children.
* children aged from 6 to 12 years old irrespective of sex.

Exclusion Criteria:

* Behavior of the child is inadequate.
* Children with dental structural defect.
* parents that refused to give informed consent.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Egyption children aged 6 to 12 years old Study group will be recruited from Abbaseya Mental Health Hospital and Advance Center For Handicapped and Autistic Children.
  Control group will be recruited from Diagnosis Clinic of Pediatric Dentistry and Dental Public Health Department at Faculty of Dentistry Cairo University.
  A selected sample will be used to select the sample for the study group and age- and gender-matched control group.
  The investigator will make an interview with the Parents of both groups, and will explain to the parents the aim of the study without any guiding to prevent any information bias may occur, then they will be assigned Informed consent, children whose parents agreed to participate in the study were recruited.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2020-11 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
occurrence of Traumatic Dental Injury | 1 year
  it will be measured by Questionnaire with binary outcome(yes/no) the investigator will make an interview with the Parents of both groups, and will explain to the parents the aim of the study without any guiding to prevent any information bias may occur.
  Traumatic childhood events are associated with a wide range of negative physical, psychological and adaptive outcomes over the life course and may lead to psychiatric illness. Autism is charactarized by repetitive, restricted behaviors and self-injury which make them vulnerable to traumatic dental injury unlike children without Autism.
  Management of Traumatic dental injuries in autistic children poses a major challenge because these children aren't have the ability to cooperate during dental care. Therefore, prevention of TDIs in ASD children is of a great importance.

SECONDARY OUTCOMES:
Risk factor of Traumatic dental injury | 1 year
  risk factor as playing activities,level of autism may contribute to traumatic dental injury.
  it will be measured by Questionnaire with binary outcome(yes/no) and scores(low/moderate/severe) the investigator will make an interview with the Parents of both groups, and will explain to the parents the aim of the study without any guiding to prevent any information bias may occur.
oral habits that contribute to TDI | 1 year
  some types of oral habits as bruxism, lip biting, thumb sucking and tongue thrusting may contribute to occurrence of traumatic dental injury Questionnaire with binary outcome(yes/no) the investigator will make an interview with the Parents of both groups, and will explain to the parents the aim of the study without any guiding to prevent any information bias may occur

CONTACTS AND LOCATIONS:
Overall Officials: marwa mousa mohamed, bachelor, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided